CLINICAL TRIAL: NCT03931408
Title: The Evaluation of Antimicrobial Bladder Instillation on the Prevalence of Chronic Urinary Tract Infections and Bladder Dysfunction in Persons With Spinal Cord Injury
Brief Title: Gentamicin Bladder Instillation in Individuals With Spinal Cord Injury Having Chronic Urinary Tract Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 18.0586
Record Dates: First submitted 2019-03-29; First posted 2019-04-30 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Neurogenic Bladder; Spinal Cord Injuries
Keywords: bladder; spinal cord injury; urinary tract infection
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Cord Injuries; Urinary Tract Infections | interventions — Gentamicins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Before the intervention, you will be randomly assigned to one of three groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Gentamicin (Experimental): Participants will be randomized into one of three groups. In this arm, participants will perform bladder instillations using a 50ml solution of gentamicin mixed with saline, 2 times per day. A formulation derived from 480 mg gentamicin sulfate diluted in 1 L normal saline will be used for instillation. Participants will be blinded during the study and will not know if they are receiving gentamicin or placebo (saline alone).
  Interventions: Drug: Gentamicin Sulfate
- Placebo instillation (saline alone) (Placebo Comparator): Participants will be randomized into one of three groups. In this arm, participants will perform bladder instillations using a 50ml solution of saline alone. Participants will be blinded during the study and will not know if they are receiving gentamicin or placebo (saline alone).
  Interventions: Other: Placebo instillation (saline alone)
- No instillation (Other): Participants will be randomized into one of three groups. In this arm participants will not receive an instillation of gentamicin or saline alone, but instead will continue standard of care. Participants will be assessed at the pre-, mid- and post-intervention time points.
  Interventions: Other: No instillation

INTERVENTIONS:
Drug: Gentamicin Sulfate — Gentamicin will be compounded for immediate use in single-dose, disposable BD 50ml Luer-Lok tip syringes. The container closure system for the diluted gentamicin sulfate solution and saline solution will be sterile and processed with depyrogenation. The solution will be slowly infused into the bladder after drainage of urine is complete. While monitoring blood pressure, the solution will remain in the participant's bladder for a least 30 minutes (unless the participant is experiencing autonomic dysreflexia, and in that case, immediately drained) with the goal of attaining 2 hours.
  Other Names: Gentamicin only
  Arms: Gentamicin
Other: Placebo instillation (saline alone) — Saline will be compounded for immediate use in single-dose, disposable BD 50ml Luer-Lok tip syringes. The container closure system for the diluted gentamicin sulfate solution and saline solution will be sterile and processed with depyrogenation. The solution will be slowly infused into the bladder after drainage of urine is complete. While monitoring blood pressure, the solution will remain in the participant's bladder for a least 30 minutes (unless the participant is experiencing autonomic dysreflexia, and in that case, immediately drained) with the goal of attaining 2 hours.
  Other Names: Saline only
  Arms: Placebo instillation (saline alone)
Other: No instillation — Participants will not receive an instillation of gentamicin or saline alone, but instead will continue standard of care. Participants will be assessed at the pre-, mid- and post-intervention time points.
  Arms: No instillation

SUMMARY:
Participants will undergo daily gentamicin bladder instillations to determine if its use will reduce the rate of symptomatic urinary tract infections (UTIs) as well as the use of oral and intravenous antibiotics in adults with chronic spinal cord injury (SCI) who have recurrent UTIs. Participants are randomized into one of three groups: 1) Gentamicin and saline instillation 2) Saline only instillation 3) Standard of care, no instillation.

DETAILED DESCRIPTION:
The purpose of this study is to determine if twice daily bladder flushing with an antibiotic solution will decrease the rate of UTIs and the use of oral medications used to treat UTIs. The occurrence of UTIs in the SCI population is high, with a rate of about 2.5 episodes per year. The inability to effectively empty the bladder increases the risk of UTIs, which are the most common medical complication after SCI. This study will help us understand the effectiveness of a local bladder therapy on preventing UTIs and improving bladder function in individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Non-progressive spinal cord injury;
* Stable medical condition;
* Bladder dysfunction as a result of spinal cord injury
* History of recurrent UTIs (defined as 3 or more within the past year or 2 or more within the past 6 months).

Exclusion Criteria:

* Signs or symptoms of serious UTI that requires the use of systemic antibiotics;
* Use of any urine-acidifying agent, bladder irrigant, or systemic antibiotic within the previous 2 weeks;
* Participants colonized with gentamicin-resistant bacteria on baseline urine culture or a gentamicin allergy/sensitivity;
* Participants with known hearing loss and/or renal disease;
* Pregnant at the time of enrollment or planning to become pregnant during the time course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Harkema, PhD, Principal Investigator — University of Louisville
Locations (1):
- Frazier Rehab, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gentamicin | Placebo Instillation (Saline Alone) | No Instillation
Started | 1 | 3 | 2
Completed | 1 | 2 | 1
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gentamicin | Placebo Instillation (Saline Alone) | No Instillation | Total
Number analyzed (Participants) | 1 | 3 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 2 | 6
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 2
  Male | 1 | 3 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 2 | 2 | 5
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Bladder Storage Using Urodynamics
Description: Assessment of Lower Urinary Tract Function: Urodynamic Bladder Compliance (mL/cm H20) based on Change in Bladder Capacity.
Time Frame: 1. Baseline (1 week) 2. Midpoint (2 months) 3. Post (4 months)
Population: Bladder Compliance
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Placebo Instillation (Saline Alone): Participants will be randomized into one of three groups. In this arm, participants will perform bladder instillations using a 50ml solution of saline alone. Participants will be blinded during the study and will not know if they are receiving gentamicin or placebo (saline alone).
  Placebo instillation (saline alone): Saline will be compounded for immediate use in single-dose, disposable BD 50ml Luer-Lok tip syringes. The container closure system for the diluted gentamicin
Arm/Group | Gentamicin | Placebo Instillation (Saline Alone) | No Instillation
Number analyzed (Participants) | 1 | 3 | 2
mL
  Baseline (1 week): number analyzed (Participants) | 1 | 3 | 1
  Baseline (1 week) | 611 | 177.67 (124.23) | 662
  Midpoint (2 months): number analyzed (Participants) | 1 | 2 | 0
  Midpoint (2 months) | 452 | 286.5 (226.98) |
  Post (4 months): number analyzed (Participants) | 0 | 2 | 0
  Post (4 months) |  | 345.5 (313.25) |

2. Secondary Outcome: Participants With Symptomatic Urinary Tract Infection
Description: number of participants with symptomatic urinary tract infection measured by the presence of Leukocyte Esterase level in urine.
Time Frame: 1. Baseline (1 week) 2. Midpoint (2 months) 3. Post (4 months)
Population: Presence of Leukocyte Esterase in Urine
Measure: Number; unit: participants
Arm/Group | Gentamicin | Placebo Instillation (Saline Alone) | No Instillation
Number analyzed (Participants) | 1 | 3 | 2
participants
  Baseline (1 week) | 1 | 3 | 2
  Midpoint (2 months): number analyzed (Participants) | 1 | 3 | 0
  Midpoint (2 months) | 1 | 3 |
  Post (4 months): number analyzed (Participants) | 0 | 3 | 0
  Post (4 months) |  | 3 |

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 6 months
Arm/Group | Gentamicin | Placebo Instillation (Saline Alone) | No Instillation
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT03931408/Prot_SAP_000.pdf